CLINICAL TRIAL: NCT06594354
Title: Examining the Effect of Oral Cryotherapy Applied to Patients Undergoing Chemotherapy on Taste Change, Appetite Level, Malnutrition Risk and Quality of Life
Brief Title: Oral Cryotherapy Applied to Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Zeynep PEHLİVAN KÖKSAL, Research Assistant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KTU-SBF-ZPK-01
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Oncologic Disease; Cancer; Chemotherapy
Keywords: Appetite; chemotherapy; malnutrition; taste dysfunction; cryotherapy; quality of life
MeSH Terms: conditions — Neoplasms; Malnutrition; Taste Disorders | interventions — Ice

STUDY DESIGN:
Intervention Model Description: Oral cryotherapy is a safe, cost-effective and easily applicable important nursing intervention used in addition to oral care in patients receiving chemotherapy, especially to prevent or reduce the severity of oral mucositis. The effectiveness of oral cryotherapy, known as the application of ice or cold water to the oral cavity, in the management of taste alteration is emphasized.
Who Masked: Care Provider
Masking Description: The data obtained from the study will be collected using a simple randomization method and a computerized randomization program will be used (www.randomizer.org). The groups determined in the program will be the intervention group and the control group; Group 1 and Group 2 will be written on two different papers and will be determined by the chemotherapy unit nurse by drawing lots. Patients who meet the sampling criteria will be divided into two randomized groups as patients who will be applied intraoral ice (intervention group) and patients who will not be applied (control group). Patients who meet the study inclusion criteria will be numbered and delivered to the researcher by the chemotherapy unit nurse on each application day. The patient will be included in the group according to the number given to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Patients in this arm will receive oral cryotherapy.The patients in the intervention group will have ice applied to their mouths for three cycles (the first cycle they met with the researcher and the second and third cycles/an average of two months) when they come for treatment at the hospital with the researcher and at home on the days they do not come for treatment, within the scope of the oral cryotherapy application protocol, they will be monitored by phone and a reminder message will be sent. During chemotherapy, ice cubes will be applied to the patients in the first hour they start receiving chemotherapy and in the same time period, three consecutive ice cubes (each ice cube melts for an average of 1.5-2 minutes/total average of 4.5-6 minutes) and the same application will be repeated three hours later. The patients will be asked to apply ice cubes at home six times (an average of 27-36 minutes/day) at two or three hour intervals for seven days, including the day they receive che
  Interventions: Other: ICE
- Control arm (No Intervention): Patients who meet the study criteria and are included in the control group will receive routine treatment and care procedures in the unit when they come to receive chemotherapy (the first cycle encountered by the researcher) and the other two cycles that follow, and will not receive oral cryotherapy.

INTERVENTIONS:
Other: ICE — The patients in the intervention group will have ice applied to their mouths for three cycles (the first cycle they met with the researcher and the second and third cycles/an average of two months) when they come for treatment at the hospital with the researcher and at home on the days they do not come for treatment, within the scope of the oral cryotherapy application protocol, they will be monitored by phone and a reminder message will be sent. During chemotherapy, ice cubes will be applied to the patients in the first hour they start receiving chemotherapy and in the same time period, three consecutive ice cubes (each ice cube melts for an average of 1.5-2 minutes/total average of 4.5-6 minutes) and the same application will be repeated three hours later. The patients will be asked to apply ice cubes at home six times (an average of 27-36 minutes/day) at two or three hour intervals for seven days, including the day they receive chemotherapy, and to record their applications on the "
  Other Names: oral ice application
  Arms: Intervention arm

SUMMARY:
Taste alteration can cause problems such as loss of appetite, inadequate energy intake and weight loss in oncology patients, increasing the risk of malnutrition and negatively affecting the quality of life of patients. It is thought that other problems mentioned can be prevented and quality of life can be improved with effective management of taste alteration. This study was planned as a randomized controlled, pre-test-post-test and experimental design to determine the effect of oral cryotherapy application on chemotherapy-induced taste alteration, thus on appetite level, malnutrition risk and quality of life.

DETAILED DESCRIPTION:
Taste changes disrupt the nutritional plan of patients, causing weight loss and an increased risk of malnutrition, and may negatively affect quality of life. However, this symptom is generally not considered life-threatening and is not considered as important or overlooked by healthcare professionals as other symptoms (nausea, vomiting, oral mucositis, pain, etc.). There is limited data in the literature regarding the management of taste changes in patients receiving chemotherapy. Studies have shown that oral cryotherapy is a method that can be used in the management of taste changes associated with chemotherapy, but more comprehensive studies are needed regarding its effectiveness.Therefore, this study was planned as a randomized controlled, pre-test-post-test and experimental design to determine the effects of oral cryotherapy on chemotherapy-induced taste changes, appetite level, malnutrition risk and quality of life.The patients included in the study will be divided into two groups by simple randomization method: patients who will receive ice cubes in the mouth (intervention/oral cryotherapy group) and patients who will not receive the application (control group).This planned study will be conducted with a total of 70 patients, 35 in the intervention group and 35 in the control group, who received treatment at the Recep Tayyip Erdoğan University Training and Research Hospital Oncology Center, Medical Oncology Department, Outpatient Chemotherapy Unit between July 2024 and July 2025 and who meet the inclusion criteria for the study.Patients who are receiving treatment in an outpatient chemotherapy unit, who can communicate verbally, who are literate, who know their diagnosis, who have an Eastern Cooperative Oncology Group (ECOG) performance score of 2 or below, who are using five chemotherapeutic agents that cause taste alteration alone or in combination (cisplatin, docetaxel, paclitaxel, oxaliplatin, vincristine), who verbally state that they have taste alteration, who do not smoke or drink alcohol or have quit, who do not use statins, hypothyroidism, antidiabetic, antipsychotic, antidepressant, hyperthyroidism, antidepressant, antihistamine, anti-inflammatory, antibiotic or antifungal medications, who do not have Chronic Kidney Disease, metabolic and liver (cirrhosis) disease and who volunteer to participate in the study will be accepted to this study.Patients whose treatment was postponed at least twice in a row, who could not be reached by phone calls, who had a World Health Organization Oral Toxicity Scale score of 1 and above, who had neutropenia (neutrophils; 1000 μL and below), who received radiotherapy to the head and neck region, who had head/neck, stomach and liver cancer, who had tooth sensitivity, who had a changed chemotherapy protocol or who were to be administered a protocol other than the specified agents, who experienced a change in taste before starting the chemotherapy protocol and who did not want to continue the study will be excluded from the study.The data of the study will be collected using the "Introductory Information Form", "ECOG Performance Scale", "World Health Organization Oral Toxicity Scale (WHOTS)", "Chemotherapy-Induced Taste Alteration Scale (C-TAS)", "Simplified Appetite Assessment Questionnaire (SNAQ)", "Malnutrition Universal Screening Tool (MUST)", "Body Mass Index Monitoring Form", "Nutritional Parameters Monitoring Form", "Oral Ice Application Record Form" and "European Organization for Research and Treatment of Cancer Quality of Life Scale (EORTC QLQ-30-Version 3.0)".Before starting the study, the scales and follow-up forms specified for the intervention (oral cryotherapy) and control groups will be filled out by the researcher in a face-to-face interview. The patients in the intervention group will be subjected to oral ice application protocol during three courses (the first course in which the researcher is seen and the second and third courses/an average of two months) at the hospital when they come for treatment, and at home on the days they do not come for treatment, and will be monitored by phone and a reminder message will be sent. During chemotherapy, ice cubes will be applied to the patients in the first hour they start receiving chemotherapy and three consecutive ice cubes (each ice cube takes an average of 1.5-2 minutes to melt/total average of 4.5-6 minutes) during the same period, and the same application will be repeated three hours later. The patients will be asked to apply ice cubes at home six times (an average of 27-36 minutes/day) at two or three-hour intervals for seven days, including the day they receive chemotherapy, and to record their applications on the "Oral Ice Application Follow-up Form".At the end of the study (approximately two months later), the scales will be re-applied to the patients in the intervention and control groups in a face-to-face interview. The pre-test and post-test data from the intervention and control groups will be collected by the researcher using a face-to-face interview technique at a time when the patients are receiving chemotherapy and are available.

ELIGIBILITY:
Inclusion Criteria:

* Those receiving treatment in an outpatient chemotherapy unit,
* Able to communicate verbally,
* Literate,
* Eastern Cooperative Oncology Group (ECOG) Performance Score of two or below,
* Knowing their diagnosis,
* Taking five chemotherapeutic agents that cause taste changes, either alone or in combination (cisplatin, docetaxel, paclitaxel, oxaliplatin, vincristine),
* Verbally stating that they experience taste changes,
* Not smoking or quitting alcohol,
* Not using statins, hypothyroidism, antidiabetic, antipsychotic, hyperthyroidism, antidepressant, antihistamine, anti-inflammatory, antibiotic and antifungal drugs,
* Not having Chronic Renal Failure (CKD), metabolic (diabetes, thyroid disease, etc.) and liver (hepatitis, cirrhosis) diseases,
* Individuals who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Patients who have had their treatment postponed at least twice in a row,
* Those with a World Health Organization Oral Toxicity Scale score of 1 and above,
* Those who have received radiotherapy to the head and neck region,
* Those with head/neck, stomach and liver cancer,
* Those who cannot be reached during phone calls,
* Those whose chemotherapy protocol has changed or who will be applied to a protocol other than the specified agents,
* Those with neutropenia (neutrophils; 1000 mcL and below),
* Those with tooth sensitivity,
* Those who have experienced a change in taste before starting the chemotherapy protocol** and
* Those who do not want to continue the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-Induced Taste Alteration Scale (C-TAS) | two months
  The scale was developed by Kano and Kanda in 2013. The scale was developed to reveal the effects of chemotherapy-induced taste changes on the individual. The validity and reliability study of the scale in Turkey was conducted by Sözeri and Kutlutürkan in 2014. In the validity and reliability study, the Cronbach alpha value of the scale was found to be 0.86. The scale consists of three subheadings, four subdimensions as "Reduction in the Perception of Basic Tastes", "Phantogeusia and Parageusia", "Discomfort" and "General Taste Changes" and a total of 18 items in a five-point Likert type (1-normal taste, 5-no taste). The scores obtained from the scale subdimensions are used in the evaluation of the scores obtained from the scale. The scores obtained from the scale subdimensions are obtained by summing up those items and dividing them by the number of items. The maximum score that can be obtained from the subdimensions and the total scale score is five, while the minimum score is one.
Simplified Nutritional Appetite Questionnaire (SNAQ) | two months
  This questionnaire, which was developed in a simple and understandable way to measure the appetite of patients, was developed by Wilson et al. in 2005 and the Cronbach alpha value was found to be 0.70. The validity and reliability of the questionnaire in Turkish was conducted by Tatar et al. in 2021 and the Cronbach alpha coefficient was found to be 0.86. The scale consists of four questions and each question has five options (a = 1 point, b = 2 points, c = 3 points, d = 4 points, e = 5 points) and is scored between 4 and 20 points in total. If the patient's score from the questionnaire is 14 points or less, this indicates that the individual is at risk for 5% weight loss in the last six months. As the total score from the questionnaire decreases, the appetite level worsens.
Malnutrition Universal Screening Tool (MUST) | two months
  It is a five-step screening method recommended by the European Society of Parenteral and Enteral Nutrition (ESPEN) and the British Association for Parenteral and Enteral Nutrition (BAPEN). The scale consists of three sections (malnutrition, malnutrition risk and obesity). Malnutrition risk is classified as low, medium and high. Scores from the categories of "Body Mass Index (BMI)", "Unexpected Body Weight Loss History" and "Acute Disease Effects" are used in the classification.
European Organization for Research and Treatment of Cancer Qıality of Life Questionnaire (EORTC QLQ-30-Version 3.0) | two months
  The EORTC QLQ-C30 was developed by the European Organization for Research and Treatment of Cancer in 1987 to assess the quality of life of cancer patients. The scale was later revised by Aaronson et al. in 1993, and the Cronbach alpha coefficient was found to be 0.70. The EORTC QLQ-C30 consists of three sub-dimensions, namely "general quality of life", "functional functions" (physical, role, cognitive, emotional, social) and "symptom scale" (fatigue, pain, nausea/vomiting, dyspnea, insomnia, anorexia, constipation, diarrhea, financial difficulties) and 30 questions. The first 28 of the scale questions are of the four-point Likert type (not at all-1; very much-4). High scores from the first 28 questions indicate low quality of life, while low scores indicate high quality of life. The 29th and 30th questions of the scale are questions that constitute the general quality of life domain.
Introductory information form | two months
  This form prepared by the researchers includes three sections. The first part includes eight questions about the sociodemographic characteristics of the patients (age, gender, marital status, employment status, etc.), the second part includes nine questions about the cancer disease and the treatment method applied (cancer type, stage, metastasis status, number of cures, chemotherapy regimen). etc.) and the third part consists of a total of 31 questions, 13 of which include questions about taste changes, appetite and malnutrition (appetite status, oral care, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep PEHLİVAN KÖKSAL, Masters, Principal Investigator — Recep Tayyip Erdogan University
Locations (3):
- Turkey (Türkiye) (3):
  - Recep Tayyip Erdogan University, Rize, Rize Province
  - Recep Tayyip Erdoğan University Training and Research Hospital, Rize, Rize Province
  - Recep Tayyip Erdoğan University, Rize, Rize Province

IPD SHARING:
Plan to Share IPD: No